CLINICAL TRIAL: NCT06070454
Title: Prospective Evaluation of Infectious Vulvovaginitis on Wound Complication Rates After Vulvar Excision for Premalignant Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Carrie Sopata, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HSR230407
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Vaginitis; Vulvar Diseases
MeSH Terms: conditions — Vaginitis; Vulvar Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Positive Perioperative Vaginitis (Experimental): Participants who test positive for BV, candida, and/or trichomonas on perioperative vaginitis swab.
  Interventions: Diagnostic Test: Vaginitis panel

INTERVENTIONS:
Diagnostic Test: Vaginitis panel — vulvovaginal swab to test for the most common causes of vulvovaginitis - bacterial vaginosis (BV), trichomonas, and candida

SUMMARY:
Primary:

* To measure the rate of perioperative vulvovaginitis in a population of patients in central VA with non-malignant vulvar disease who require surgical excision
* To correlate the rate of vulvovaginitis with rate of wound cellulitis and incisional breakdown in patients undergoing SPV/WLE for vulvar disease We will use a vulvovaginal swab to test for the most common causes of vulvovaginitis - bacterial vaginosis (BV), trichomonas, and candida. The swab will be collected preoperatively on day of surgery. The outcome will be evaluated by phone call to patient at 1 week after surgery and physical exam at the postoperative visit between 4-6 weeks.

DETAILED DESCRIPTION:
Primary:

* To measure the rate of perioperative vulvovaginitis in a population of patients in central VA with non-malignant vulvar disease who require surgical excision
* To correlate the rate of vulvovaginitis with rate of wound cellulitis and incisional breakdown in patients undergoing SPV/WLE for vulvar disease We will use a vulvovaginal swab to test for the most common causes of vulvovaginitis - bacterial vaginosis (BV), trichomonas, and candida. The swab will be collected preoperatively on day of surgery. The outcome will be evaluated by phone call to patient at 1 week after surgery and physical exam at the postoperative visit between 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age
* Has histologically confirmed non-malignant vulvar pathology
* Is scheduled or planning for WLE/SPV
* Signed informed consent obtained prior to any protocol specific procedures

Exclusion Criteria:

* Unable to give informed consent
* Women who are pregnant or nursing (lactating) women at time of consent
* No prior RT
* No recent antibiotic use within the last 3 weeks or 5.5 times the half-life of the antibiotic (whichever is shorter)
* No history of prior malignancy within the last 3 years that required systemic chemotherapy or radiation
* Not immunosuppressed or compromised
* No active HIV (must have undetectable viral load)
* Chronic treatment with corticosteroids or other immunosuppressive agents including topical corticosteroids in the pelvis. Inhaled corticosteroids are allowed
* No active uncontrolled severe infections (not responding to antibiotics), except acute or chronic pelvic inflammatory disease
* Uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
the rate of perioperative vulvovaginitis | 8 weeks
  To measure the rate of perioperative vulvovaginitis in a population of patients in central VA with non-malignant vulvar disease who require surgical excision
rate of vulvovaginitis with rate of wound cellulitis and incisional breakdown | 8 weeks
  To correlate the rate of vulvovaginitis with rate of wound cellulitis and incisional breakdown in patients undergoing SPV/WLE for vulvar disease

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No